CLINICAL TRIAL: NCT07172633
Title: Effects of Scenario-Based Simulation Teaching Combined With Virtual Technology on Knowledge, Empathy, and Communication and Assessment Skills in Dementia Care Among Nursing Students
Brief Title: Effects of Dementia Scenario-Based Simulation Teaching Combined With Virtual Technology Among Nursing Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huei-Chuan Sung (Other)
Responsible Party: Sponsor-Investigator, Huei-Chuan Sung, Associate professor, Tzu Chi University
Organization: Tzu Chi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PMN1141602
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Dementia Simulation-based Teaching
Keywords: Simulation-based teaching; virtual technology; dementia; nursing student
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data assessors will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scenario-based simulation teaching with virtual technology (Experimental): 5-week scenario-based simulation teaching with a virtual coach intervention in addition to regular dementia care lectures
  Interventions: Other: scenario-based simulation teaching with virtual technology
- traditional dementia case discussions (Active Comparator): 5-week traditional dementia case discussions in addition to regular dementia care lectures
  Interventions: Other: traditional dementia case discussions

INTERVENTIONS:
Other: scenario-based simulation teaching with virtual technology — 5-week scenario-based simulation teaching with a virtual coach acting as an older adult with dementia in addition to regular dementia care lectures
  Arms: Scenario-based simulation teaching with virtual technology
Other: traditional dementia case discussions — 5-week traditional dementia case discussions in addition to regular dementia care lectures
  Arms: traditional dementia case discussions

SUMMARY:
This study aims to evaluate the effects of scenario-based simulation teaching with virtual technology on dementia knowledge, empathy, communication, and assessment skills among nursing students.

DETAILED DESCRIPTION:
This two-group randomised controlled trial aims to evaluate the effects of scenario-based simulation teaching with virtual technology on dementia knowledge, empathy, communication, and assessment skills among nursing students.

The interventional group will receive the 5-week scenario-based simulation teaching with a virtual coach in addition to regular dementia care lectures.

The control group will receive the 5-week traditional dementia case discussions in addition to regular dementia care lectures.

Both groups will be assessed for their dementia knowledge, empathy, communication, and assessment skills at baseline, week 12, and week 18.

ELIGIBILITY:
Inclusion Criteria:

* college nursing students with ages ranging from 18 to 40 years,
* Taiwanese nationality,
* provide informed consent to participate in the study.

Exclusion Criteria:

* college nursing students who do not meet the inclusion criteria

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Dementia Knowledge Assessment Scale | baseline, week 12, week 18
  Dementia Knowledge
Jefferson Scale of Empathy | baseine, week 12, week 18
  empathy
Nursing Students' Communication Behavior with Dementia Patients Scale | baseine, week 12, week 18
  Communication behavior with dementia patients
Health Professionals Communication Skills Scale | baseline, week 12, week 18
  communication skills

SECONDARY OUTCOMES:
Dementia Assessment Practice Rubrics | baseline, week 12, week 18
  assessment skills for people with dementia

CONTACTS AND LOCATIONS:
Locations (1):
- Tzu Chi University, Hualien City, Hualien, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided